CLINICAL TRIAL: NCT02035878
Title: Probiotics and the Microbiome: Clinical Intervention Trial for Anxiety and Depression
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Acadia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: POTTERHUNTER_PROBIOTICS_2013
Record Dates: First submitted 2014-01-08; First posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Anxiety; Depression
Keywords: anxiety; depression; probiotics; adult; human; depression anxiety stress scale; anxiety sensitivity index
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics (Active Comparator): 400mg probiotic capsule taken once daily for ten weeks
  Interventions: Other: Probiotics
- Placebo (rice flour) (Placebo Comparator): 400mg placebo capsule containing rice flour taken once daily for ten weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Other: Probiotics — probiotic intervention: 400mg of probiotic capsule
  Other Names: Organic Probiotics 7 Strains 20 Billion per gram
  Arms: Probiotics
Drug: Placebo — placebo comparator
  Other Names: 400 mg white rice flour capsules
  Arms: Placebo (rice flour)

SUMMARY:
The proposed project will investigate the effects of probiotics on anxiety and associated psychological and physiological factors in humans. The therapeutic potential of probiotics for reducing anxiety and other factors associated with a disrupted microbiome will be assessed in a double-blind placebo-crossover design. Based on the research findings to date, it is hypothesized that probiotics will reduce anxiety and depressive symptoms.

DETAILED DESCRIPTION:
Purpose

The human microbiome, also known as microflora, is comprised of the bacterial colonies of the body. Although bacteria are commonly associated with illness, there are good bacteria known as probiotic bacteria that grow naturally in the microbiome of the human gut. Probiotic bacteria are live microorganisms and consist of approximately 400 different bacterial strains that support life in their host organism. The gut microbiome, also known as intestinal flora, plays a role in normal human development, digestion, body weight, nutrition, and immune system regulation, in addition to influencing various neurological functions. It has been found that environmental factors including antibiotics, illness, stress, and diet can alter an individual's microbiome through their effects on probiotic bacteria situated in the gut microflora.

Although probiotic bacteria grow naturally in the human gut, acquisition of the gut microbiome varies in each individual depending on various factors, including birth method and early diet. Research suggests that newborns' first exposure to bacteria and acquisition of the first components of their microbiome takes place during birth. Infants acquire their mothers' bacteria as they pass through the vaginal canal during childbirth. Research indicates that, for this reason, children born through cesarean section have a less diverse microbiome (Dominguez-Bello, Costello, Contreras, Magris, Hidalgo, Fierer, & Knight, 2010). Research also suggests that following birth, infants continue to acquire their gut microbiome in the first two years of life under the influence of dietary nutrition. For example, in a study of six breast-fed and six formula fed infants, those who consumed a specially enriched formula that contained both prebiotics (substances that feed probiotics) and a variety of probiotic bacteria had a much more diverse intestinal flora than those who received breast milk (Harmsen, Wildeboer-Veloo, Raangs, Wagendorp, Klijn, Bindels, & Welling, 2000). Please note that this study does not negate the benefits of breast milk and was intended to assess the effect of heightened prebiotic and probiotic concentrations in a baby formula that was chemically similar to breast milk.

Because probiotic bacteria are acquired naturally from environmental sources in addition to growing normally in the human body, it is safe for humans to consume probiotics. Furthermore, Health Canada has labeled probiotics a natural health product (NHP) safe for human consumption. Common foods we eat each day contain probiotic bacteria that enrich our intestinal flora. For example, yogurt and cheese contain probiotic bacteria. There has been a recent upsurge in interest on probiotics amongst researchers as the positive effects of probiotics on the gut microbiome and recognition of their great therapeutic potential for a wide variety of conditions increases.

The Microbiome and Physical Health

Research has shown that probiotic bacterial strains, such as Bifidobacteria and Lactobacilli, aid in the treatment of Irritable Bowel Syndrome and other gastrointestinal and bowel diseases by inhibiting the colonization and growth of bacteria that cause disease. In addition, the gut microbiome is believed to play an integral role in regulating healthy immune system functioning. Immune system functioning is maintained by homeostatic relationships with the microbiome, which in turn plays a role in the development of lymphoid tissues and the immune system (Hooper, Littman, & Macpherson, 2012). Imbalances in gut microflora have been associated with impaired immune responses.

The Microbiome and Mental Health

The microbiome has been associated with a variety of mental health conditions. Researchers have dubbed this connection "the gut-brain axis" (Forsythe, Sudo, Dinan, Taylor, & Bienenstock, 2010). Bacteria in the gut have been found to produce GABA and serotonin, although the exact mechanism by which these gastrointestinally produced neurotransmitters influence brain functioning is unknown at this time. However, disruptions in the microbiome have been associated with autism, as well as with anxiety and depressive disorders.

Imbalances in the intestinal flora as a result of early antibiotic use, for example, have also been implicated in the development of autism. Probiotics have been shown to aid in the treatment of autistic symptoms by promoting the growth of beneficial bacteria and inhibiting the growth of harmful bacteria. Researchers have identified an overgrowth of certain strains of Clostridia that produce propionic acid in the guts of autistic children. Propionic acid is a neurotoxin that crosses the blood-brain barrier and could disrupt normal brain development in early childhood (Parracho, Gibson, Knott, Bosscher, Kleerebezem, & McCartney, 2010).

Disruptions in the development of normal microflora have also been associated with alterations in stress reactivity that continue into later life. For example, various metabolic pathways, such as those involving bile acids and steroid hormone synthesizers, that are necessary for bodily functions depend on a healthy microbiome (Antunes, Han, Ferreira, Lolic, Borchers, & Finlay, 2011). Research shows that antibiotic use early in life leads to a reduction in intestinal flora and diversity and may be involved in causing a physiological state of alert, akin to a trait known as "anxiety sensitivity". Anxiety sensitivity refers to a tendency in some individuals to monitor their physiological state continuously and misinterpret normal fluctuations in homeostasis as life threatening events. In animal studies, consumption of probiotics leads to reductions in anxiety-related behaviours as well as alterations in the GABA receptors that mediate stress-related hormones (Bravo, Forsythe, Chew, Escaravage, Savignac, Dinan, Bienenstock, & Cryan, 2011). The beneficial effects of gut microbiota on stress and anxiety have also been evidenced when comparing germ-free mice (i.e., mice with no microbiome) to mice with rich intestinal microflora. Mice with rich intestinal microflora show less stress reactivity than germ-free mice.

Current Proposal

The proposed project will investigate the effects of probiotics on anxiety and associated psychological and physiological factors in humans. The therapeutic potential of probiotics for reducing anxiety and other factors associated with a disrupted microbiome will be assessed in a double-blind placebo-crossover design. Based on the research findings to date, it is hypothesized that probiotics will reduce anxiety and depressive symptoms.

Methodology

Seventy-five male and female participants over the age of 18 years will be recruited through advertisements posted in various locations around the Wolfville area, as well as local newspapers and social media sites such as Facebook. Online advertisements including a link to a website containing information about study eligibility and requirements (http://www.probioticstudy.com) will be posted on the Facebook groups of various organizations in Wolfville, including Inner Sun Yoga Center, Wolfville Farmer's Market, and EOS Fine Foods community board, as well as in local newspapers such as the Grapevine and the Advertiser (see Appendix A). Information brochures will be distributed to the Valley Regional Hospital, Eastern Kings Memorial Health Centre, and Mud Creek Medical Co-op Ltd. for display in their waiting rooms (see Appendix B). Advertisement posters will also be posted in the Wolfville area (including the Acadia Athletic Complex community board, Wolfville Shopper's Drug Mart, and Wolfville Post Office community board) with pull-tabs containing the website URL for the study information page (see Appendix C). An all-staff email will also be sent to Acadia University staff targeted at non-academic occupations for recruitment (see Appendix D).

Because there is limited research on participants under the age of 18, participants must be at least 18 years of age. Participants must also live within driving distance of Wolfville, Nova Scotia, be able to come to Wolfville for appointments with the researchers, and have a valid email address. Exclusionary criteria for participation include having an academic-related occupation, including University/College professor or student (to avoid cohort effects related to specific fluctuations in conditions associated with high stress during the academic term); having HIV/AIDS; currently undergoing chemotherapy; having a diagnosed serious metabolic, immune, or digestive problem, including cancer, Crone's disease or ulcerative colitis, multiple sclerosis, lupus, Addison's disease or other form of adrenal insufficiency; currently using medication for anxiety; taking probiotic capsules; taking antibiotics; or having any other serious medical illness.

Once potential participants have reviewed the information on the study website and indicated that they wish to participate, they will be directed to an informed consent page. By checking the box and clicking "Submit" on the online informed consent page, they will indicate their consent to participate and will be directed to a demographic questionnaire (see Appendix E). The questionnaire will contain questions about the participants' health, medical history, and foods they consume. All data collected online during this study will be housed on a Canadian server to avoid Patriot Act issues associated with data housed on U.S. servers. The researcher will schedule appointments with participants who give online consent to participate.

The study will be carried out over a 22-week period, during which the participants will consume an oral probiotic for 10 weeks and a placebo (an inert substance with no therapeutic effect) for 10 weeks, with a two-week washout period in between. Participants will receive either the probiotic or the placebo for the first ten weeks and the other for the second 10 weeks. Neither the participant nor the researcher administering the probiotics and placebos will be aware which one the participant is taking. Because this a double-blind design, only the supervisor, Dr. Susan Potter, will be privy to the experimental condition of the participants. The supervisor will randomly assign participants to either a placebo or probiotic condition.

The probiotic used in this study will be Organic Probiotics 7 Strains 20 Billion per gram purchased from Prescribed For Life. This is a natural organic probiotic powder including Acidophilus, Bifidum, Casei, and Rhamnosus strains of probiotic bacteria, 400mg per capsule. Placebo capsules will contain 400mg of rice flour. Each participant will receive two pill bottles - one with 70 probiotic capsules for ten weeks and another with 70 placebo capsules for ten weeks. These capsules are to be consumed orally, one capsule per day.

The researcher and supervisor will schedule a meeting with each participant to provide detailed instructions for the study and to obtain informed consent for each participant's continuation in the study (see Appendix F and Appendix G). At the initial appointment, the ten-week appointment, and the final twenty-week appointment, participants will complete the Depression Anxiety and Stress scale (DASS) and the Anxiety Sensitivity Index (ASI). Participants will complete these measures three times during the study period in order for the researchers to measure change in anxiety and depression symptoms across the three time points. At each of these meetings participants will also be given their bottle of either probiotics capsules or placebo capsules to be taken over the 10-week period. At their ten-week appointment, participants will also be given copies of the DASS and ASI to be completed at the end of the study (see Appendix H). At the third and final appointment, participants will bring in their completed questionnaires and be given the opportunity to ask any questions they may have about the study, as well as complete a ballot for the prize draws. If they wish to know during which phases they received the probiotic and placebo capsules, they will be told that the information will be emailed to them once the study is complete.

Participants will be contacted by the researcher on the third and sixth day of each phase (probiotic and placebo) via email to check in and answer any questions they may have (see Appendix I). Participants will be asked to complete a brief questionnaire once every two weeks during the study period, which should take no longer than 5 minutes to complete (see Appendix J and Appendix K), to chart any changes in anxiety and/or physical health, as well as to keep the lines of communication open should any questions arise.

Consent

Participants will complete two consent forms, one online prior to the collection of demographic and identifying information and one prior to commencing the probiotic phase of the study (see Appendix E, and Appendix G, respectively).

Deception and Debriefing

Although not technically deception, participants will receive either a placebo or probiotic for ten-week intervals in the study period but will not be told which of the two they are receiving, although they will be informed that they will not be told. Upon completion of the study, participants who wish to know will be told which of the two (probiotics or placebo) they received during each ten-week period. Participants will also be given the opportunity to have all of their questions answered by the researcher and those who wish to receive a copy of the results will be sent them via email once the study is complete.

Risks and Benefits

Probiotics are good bacteria that grow naturally in the human gut. To date, there are no published risks associated with probiotic consumption. Nevertheless, participants will be contacted twice during the first week of each phase (probiotic and placebo) to ensure they are not experiencing any adverse side effects. In addition, participants will submit updates on their physical and mental health every two weeks throughout the study in addition to being encouraged to contact the researchers should they have any concerns during the study period.

It is possible that participants may be made more aware of any anxious or depressive symptoms they are experiencing through participation in this research project and, as a result of increased attending, may experience increases in their emotional distress. To address these concerns, participants will be provided with specific contact information for mental health service providers in the Wolfville area.

Although direct benefits to the participants are uncertain at this point, it is possible that they may experience a reduction in anxiety and/or depressive symptoms, and it is quite likely they will experience a reduction in any physiological bowel-related symptoms, as a result of taking the probiotics. However, it will be impossible to determine if any improvements in symptoms are attributable to the probiotic intervention until the study is complete.

Confidentiality

Confidentiality will be maintained at all times. Once they are enrolled in the study, each participant will be assigned a unique code number that will be used on all questionnaires and other data. Participants' names will not appear in conjunction with any data except for the initial online questionnaire. Once potential participants have been contacted about their participation in the intervention phase of the study, the online questionnaire data will be removed from the server and names will be replaced with code numbers. A master list of code numbers and names will be kept in a password-protected file in a separate folder on the researcher's password-protected computer.

Data Security: All paper questionnaires will be stored in a locked filing cabinet in a locked office. All electronic data files will be stored on a password-protected computer. Because this area of research is relatively new, data will be kept indefinitely as it may help to guide future studies.

ELIGIBILITY:
Inclusion Criteria:

* I have a valid email address that I check routinely and daily access to the internet.
* I experience symptoms of anxiety and/or depression.
* I am over the age of 18.
* I am within driving distance of Wolfville, Kingston-Greenwood, or Halifax, Nova Scotia, and would be able to come to Wolfville or Halifax for appointments with the researchers. OR I am not within driving distance of Wolfville, Nova Scotia or Halifax Nova Scotia, but am a resident of Canada and would be available for telephone or online conference calls.

Exclusion Criteria:

* I am a University/College professor or student.
* I have one or more of the following diagnosed conditions: Cancer, Crohn's disease or ulcerative colitis, Multiple sclerosis, Lupus, Addison's Disease or other form of adrenal insufficiency
* I am currently taking antibiotics or probiotic capsules.*
* I have diagnosed HIV/AIDS.
* I am currently undergoing chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-08; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Depression Anxiety and Stress Scale (DASS) - Time 1 (we are assessing change over time) | Baseline (at first meeting)
  A self-report questionnaire that assesses current symptoms of depression, anxiety, and feelings related to stress. Note that this measure is completed by participants at three different time points in order to assess change in symptoms across time points.
Depression Anxiety and Stress Scale (DASS) - Time 2 (we are assessing change over time) | administered at 10 weeks
  A self-report questionnaire that assesses current symptoms of depression, anxiety, and feelings related to stress. Note that this measure is completed by participants at three different time points in order to assess change in symptoms across time points.
Depression Anxiety and Stress Scale (DASS) - Time 3 (we are assessing change over time) | Administered at 22 weeks (i.e., the end of the study)
  A self-report questionnaire that assesses current symptoms of depression, anxiety, and feelings related to stress. Note that this measure is completed by participants at three different time points in order to assess change in symptoms across time points.
Anxiety Sensitivity Index (ASI) - Time 1 (we are assessing change over time) | Baseline (at first meeting)
  A self-report questionnaire that assesses anxiety sensitivity -- the degree to which an individual focuses on and notices (and avoids) physical changes related to anxiety. Note that this measure is completed by participants at three different time points in order to assess change in anxiety sensitivity across time points.
Anxiety Sensitivity Index (ASI) - Time 2 (we are assessing change over time) | administered at 10 weeks
  A self-report questionnaire that assesses anxiety sensitivity -- the degree to which an individual focuses on and notices (and avoids) physical changes related to anxiety. Note that this measure is completed by participants at three different time points in order to assess change in anxiety sensitivity across time points.
Anxiety Sensitivity Index (ASI) - Time 3 (we are assessing change over time) | administered at 22 weeks
  A self-report questionnaire that assesses anxiety sensitivity -- the degree to which an individual focuses on and notices (and avoids) physical changes related to anxiety. Note that this measure is completed by participants at three different time points in order to assess change in anxiety sensitivity across time points.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Susan Potter, PhD, Principal Investigator — Acadia University
Locations (1):
- Acadia University, Wolfville, Nova Scotia, Canada

REFERENCES:
- [Background] Dominguez-Bello MG, Costello EK, Contreras M, Magris M, Hidalgo G, Fierer N, Knight R. Delivery mode shapes the acquisition and structure of the initial microbiota across multiple body habitats in newborns. Proc Natl Acad Sci U S A. 2010 Jun 29;107(26):11971-5. doi: 10.1073/pnas.1002601107. Epub 2010 Jun 21. PMID 20566857
- [Background] Harmsen HJ, Wildeboer-Veloo AC, Raangs GC, Wagendorp AA, Klijn N, Bindels JG, Welling GW. Analysis of intestinal flora development in breast-fed and formula-fed infants by using molecular identification and detection methods. J Pediatr Gastroenterol Nutr. 2000 Jan;30(1):61-7. doi: 10.1097/00005176-200001000-00019. PMID 10630441
- [Background] Hooper LV, Littman DR, Macpherson AJ. Interactions between the microbiota and the immune system. Science. 2012 Jun 8;336(6086):1268-73. doi: 10.1126/science.1223490. Epub 2012 Jun 6. PMID 22674334
- [Background] Forsythe P, Sudo N, Dinan T, Taylor VH, Bienenstock J. Mood and gut feelings. Brain Behav Immun. 2010 Jan;24(1):9-16. doi: 10.1016/j.bbi.2009.05.058. Epub 2009 May 28. PMID 19481599
- [Background] Bienenstock J. Commensal communication to the brain: pathways and behavioral consequences. Microb Ecol Health Dis. 2012 Aug 24;23. doi: 10.3402/mehd.v23i0.19007. eCollection 2012. No abstract available. PMID 23990826
- [Background] Bravo JA, Forsythe P, Chew MV, Escaravage E, Savignac HM, Dinan TG, Bienenstock J, Cryan JF. Ingestion of Lactobacillus strain regulates emotional behavior and central GABA receptor expression in a mouse via the vagus nerve. Proc Natl Acad Sci U S A. 2011 Sep 20;108(38):16050-5. doi: 10.1073/pnas.1102999108. Epub 2011 Aug 29. PMID 21876150
- [Background] Antunes LC, Han J, Ferreira RB, Lolic P, Borchers CH, Finlay BB. Effect of antibiotic treatment on the intestinal metabolome. Antimicrob Agents Chemother. 2011 Apr;55(4):1494-503. doi: 10.1128/AAC.01664-10. Epub 2011 Jan 31. PMID 21282433